CLINICAL TRIAL: NCT03568188
Title: Phase 2, Multicenter, Prospective Cohort Study, Estimating the Efficacy of Focused HIFU Therapy in Patients With Localized Intermediate Risk Prostate Cancer
Brief Title: Efficacy Evaluation of Focused HIFU (High Intensity Focused Ultrasound) Therapy in Patients With Localized Intermediate Risk Prostate Cancer
Acronym: FOCALE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0292; 2018-A01171-54 (Other: ID-RCB)
Record Dates: First submitted 2018-06-06; First posted 2018-06-26 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; HIFU focal; adverse effect; intermediate risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Therapeutics; Surveys and Questionnaires; Hematologic Tests; Urinalysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU treatment (Experimental): 170 patients with prostate cancer of intermediate risk receive the immediate treatment with focal HIFU. The treatment area will be defined using MRI data and 3D biopsies. A safety distance of at least 9 mm will be defined around the tumor. An intraoperative contrast echocardiographic control will be performed to evaluate the necrotic area. If necessary, additional HIFU lesions will be performed during the same session. In case of residual tumor demonstrated during control biopsies, additional treatment of this tumor with focal HIFU may be proposed. Patients will also have PSA (Prostate-Specific Antigen) dosage, MRI (Magnetic Resonance Imaging) exam, questionnaires and prostatic biopsies during their follow up. If the patient decides to participate in the ancillary study, a blood test (for immunological analyzes and detection of CTC (circulating tumor cells)) and a urine test (for PCA3 (The prostate cancer antigen 3 gene) test) will be performed during their follow up.
  Interventions: Procedure: treatment with focal HIFU; Biological: PSA dosage; Device: MRI; Other: Questionnaires; Procedure: Prostatic biopsies; Biological: blood test; Biological: urine test

INTERVENTIONS:
Procedure: treatment with focal HIFU — HIFU treatment will be conducted with the Focal One® device. The treatment area will be defined using MRI data and 3D biopsies. A safety distance of at least 9 mm will be defined around the tumor. An intraoperative contrast echocardiographic control will be performed to evaluate the necrotic area. If necessary, additional HIFU lesions will be performed during the same session. In case of residual tumor demonstrated during control biopsies, additional treatment of this tumor with focal HIFU may be proposed.
Biological: PSA dosage — PSA dosage will be regularly performed during patient follow up thanks to blood sampling.
Device: MRI — MRI exam will be regularly performed during patient follow up.
Other: Questionnaires — Patients will have to complete five questionnaires during their follow up : QLQ-C30 (Quality of Life questionnaire), EPIC-26 (The Expanded Prostate Cancer Index Composite), IPSS (International Prostate Score Symptom), IIEF-5 (The International Index of Erectile Function).
Procedure: Prostatic biopsies — Prostatic biopsies will be regularly performed during patient follow up.
Biological: blood test — if the patient decides to participate in the ancillary study, a blood test (for immunological analyzes and detection of CTC (circulating tumor cells)) will be performed during their follow up.
Biological: urine test — if the patient decides to participate in the ancillary study, a urine test (for PCA3 test) will be performed during their follow up.

SUMMARY:
The aim of the focal treatment HIFU is to destroy the cancer without causing side effects in contrast to radical treatments. Radical treatments (surgery or radiation therapy) are the standard therapies for patient with intermediate risk localized prostate cancer and good life expectancy (prostatectomy if life expectancy10 years) By destroying only the part of the gland that harbors cancer, it may indeed be possible to provide efficient cure of the disease while minimizing treatment-induced morbidity (incontinence and loss of potency). Around 20% of patients presented with a unilateral tumor: this patients are currently treated radically. No study published papers reported outcomes of a large population (>100) with intermediate risk cancers treated with Focal-HIFU (conducted with the Focal One® device). Focal therapy must be only offer within clinical trial setting (EAU (European Association of Urology) Guidelines ). The aim of this cohort will be to determine the success rate of Focal-HIFU in this intermediate risk population. The result the study will be used for calculation the arms of a future random study

ELIGIBILITY:
Inclusion Criteria:

* Patient having been clearly informed of the study and having accepted, with sufficient reflection time, to participate by signing the informed consent form of the study.
* Age between 50 and 80 years with a life expectancy of more than 5 years. Patients between the ages of 75 and 80 will need to have a G8 score > 14.
* Initial diagnosis of localized prostate cancer (T1c or T2a) with the following characteristics:

  * A multiparametric MRI showing a single invasive tumor focus at most two contiguous sextants confirmed by biopsies (index tumor). Patients with multiple suspected MRI foci may be included if only one of these foci is confirmed by targeted biopsies.
  * Gleason score= 7 (3+4).
  * Tumor accessible to a Focal-HIFU treatment. For apical tumor, it must be localized more than 9 mm from the external sphincter
* PSA ≤ 15ng / ml.
* Patient affiliated with health insurance or beneficiary of an equivalent plan.

Exclusion Criteria:

* Contraindications to treatment with HIFU-F:

  * Tumor not accessible.
  * Multiple intra prostatic calcifications inducing, on ultrasound, a shadow cone in the prostate preventing the penetration of ultrasound and thus the realization of the treatment.
  * History of pelvic irradiation
  * Presence of an implant (stent, catheter) located less than 1 cm from the treatment area.
  * Fistula of the urinary tract or rectum.
  * Anal or rectal fibrosis, anal or rectal stenosis or other abnormalities making it difficult to insert the Focal One® probe.
  * Anatomical abnormality of the rectum or rectal mucosa.
  * Patient with artificial sphincter, penile prosthesis or intra prostatic implant, eg stent.
  * History of intestinal inflammatory pathology.
  * Uro-genital infection in progress (the infection to be treated before HIFU treatment).
  * Anterior surgery at the level of the anus or rectum making the introduction of the probe impossible.
  * Allergy to latex.
  * Thickness of the rectal wall> 10mm.
* TURP indication. Bladder neck incision is allowed.
* Patient with a medical contraindication to Sonovue® injection.
* Patient with a medical contraindication on MRI.
* Patient already treated for prostate cancer (hormone therapy, radiotherapy, surgery).
* History of uncontrolled cancer and / or treated for less than 5 years (with the exception of basal cell skin cancer).
* History of pelvic radiotherapy.
* History of sclerosis of the bladder neck or urethral stenosis.
* Patient with a several bleeding risk according to medical advice (patient with oral anticoagulant therapy must receive an alternative therapy).
* Patients with unstable neurological pathology.
* Patient who has been treated for a therapeutic trial within 30 days of enrollment or who wishes to participate in an ongoing study that may interfere with this study.
* Legal person protected by law.
* Patient not able to understand the objectives of the study or refusing to comply with postoperative instructions.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
patient proportion with controlled disease (Control of the pathology) | 12 months
  The main objective is the estimation of FOCAL HIFU treatment efficacy defined as the percentage of positive biopsies in the treated lobe at 12 months after inclusion.

SECONDARY OUTCOMES:
proportion of patients needing additional treatment | 12 months
  The objective is to determine the proportion of patients needing additional treatment (focal or radical) at 12 months. This includes patients who wish or require radical treatment (prostatectomy, radiotherapy), total focal treatment, or additional focal treatment.
proportion of patients needing additional treatment | 48 months
  The objective is to determine the proportion of patients needing additional treatment (focal or radical) at 48 months. This includes patients who wish or require radical treatment (prostatectomy, radiotherapy), total focal treatment, or additional focal treatment.
proportion of patients needing additional radical treatment | 12 months
  The objective is to determine the proportion of patients needing additional radical treatment at 12 months. This includes patients who wish or require prostatectomy or radiotherapy total focal treatment.
proportion of patients needing additional radical treatment | 48 months
  The objective is to determine the proportion of patients needing additional radical treatment at 48 months. This includes patients who wish or require prostatectomy or radiotherapy total focal treatment.
rate of positive biopsies | 12 months
  The rate of positive biopsies in the untreated lobe and treated lobe evaluated and will be used to evaluate the carcinologic evolution at 12 months.
rate of positive biopsies | 24 months
  The rate of positive biopsies in the untreated lobe and treated lobe evaluated and will be used to evaluate the carcinologic evolution at 24 months.
rate of positive biopsies | 48 months
  The rate of positive biopsies in the untreated lobe and treated lobe evaluated and will be used to evaluate the carcinologic evolution at 48 months.
clinically significant cancer rate | 48 months
  The clinically significant cancer rate (Gleason 7 or invasion of more than 3 biopsies or invasion> 3 mm regardless of Gleason) in the untreated lobe and the treated lobe will be measured and will be used to evaluate the carcinologic evolution at 48 months.
Gleason score | 12 months
  Evolution of the Gleason score (appearance of Gleason ≥7) will be measured and will be used to evaluate the carcinologic evolution at 12 month.
  The Gleason score is a prognosis factor for prostate cancer. It is based prostate cancer cells architecture from biopsies. The more the architectures of prostate cancer cell is destroyed, the worse is the prognosis. The score grades from 3 to 5, 5 being the more destroyed, the score 1 and 2 being normal cells. When there is more than one tumor cells population in the prostate, the score is composed of the sum of the most 2 frequents grade. For example a Gleason 7 tumor could be 3+4 or 4+3, the 4+3 being more aggressive.
Gleason score | 24 months
  Evolution of the Gleason score (appearance of Gleason ≥7) will be measured and will be used to evaluate the carcinologic evolution at 24 month.
  The Gleason score is a prognosis factor for prostate cancer. It is based prostate cancer cells architecture from biopsies. The more the architectures of prostate cancer cell is destroyed, the worse is the prognosis. The score grades from 3 to 5, 5 being the more destroyed, the score 1 and 2 being normal cells. When there is more than one tumor cells population in the prostate, the score is composed of the sum of the most 2 frequents grade. For example a Gleason 7 tumor could be 3+4 or 4+3, the 4+3 being more aggressive.
Gleason score | 48 months
  Evolution of the Gleason score (appearance of Gleason ≥7) will be measured and will be used to evaluate the carcinologic evolution at 48 month.
  The Gleason score is a prognosis factor for prostate cancer. It is based prostate cancer cells architecture from biopsies. The more the architectures of prostate cancer cell is destroyed, the worse is the prognosis. The score grades from 3 to 5, 5 being the more destroyed, the score 1 and 2 being normal cells. When there is more than one tumor cells population in the prostate, the score is composed of the sum of the most 2 frequents grade. For example a Gleason 7 tumor could be 3+4 or 4+3, the 4+3 being more aggressive.
Appearance of another cancerous focus in the other half of the prostate | 12 months
  Appearance of another cancerous focus in the other half of the prostate will be supervised and will be used to evaluate the carcinologic evolution at 12 months.
Appearance of another cancerous focus in the other half of the prostate | 24 months
  Appearance of another cancerous focus in the other half of the prostate will be supervised and will be used to evaluate the carcinologic evolution at 24 months.
Appearance of another cancerous focus in the other half of the prostate | 48 months
  Appearance of another cancerous focus in the other half of the prostate will be supervised and will be used to evaluate the carcinologic evolution at 48 months.
Appearance of metastases | 12 months
  Appearance of metastases (lymph node or bone) will be supervised and will be used to evaluate the carcinologic evolution at 12 months.
Appearance of metastases | 24 months
  Appearance of metastases (lymph node or bone) will be supervised and will be used to evaluate the carcinologic evolution at 24 months.
Appearance of metastases | 48 months
  Appearance of metastases (lymph node or bone) will be supervised and will be used to evaluate the carcinologic evolution at 48 months.
Appearance of an extra capsular extension | 12 months
  Appearance of an extra capsular extension will be supervised and will be used to evaluate the carcinologic evolution at 12 months.
Appearance of an extra capsular extension | 24 months
  Appearance of an extra capsular extension will be supervised and will be used to evaluate the carcinologic evolution at 24 months.
Appearance of an extra capsular extension | 48 months
  Appearance of an extra capsular extension will be supervised and will be used to evaluate the carcinologic evolution at 48 months.
Overall survival | 48 months
  Overall survival at 48 months will be measured from the date of inclusion to the date of death, all causes of death combined or the date of last new or point date to 48 months.
Prostate cancer specific survival | 48 months
  Prostate cancer specific survival at 48 months will be measured from the date of inclusion to the date of death related to prostate cancer or the date of last new or point date to 48 months
Recurrence free survival | 48 months
  Prostate cancer specific survival at 48 months will be measured from the date of inclusion to the date of first metastasis , or the date of last new or point date to 48 months.
Proportion of serious adverse effect | 48 months
  comparison of the proposition of serious adverse effect at 48 months
Quality of life score | over the 48 months
  quality of life will be assessed using the QLQC30 (Quality of Life questionnaire) questionnaire.
  It is a specific questionnaire to determine the quality of life a patient with cancer. It is composed of 30 questions with 4 potential answers going from: not at all, a little, enough or a lot, within 28 questions and with a visual scale going from 1 to 7 (7 being excellent and 1 being very bad) for the last 2 questions. The raw score is established by adding the score of each question and a linear transformation range it from 0 to 100. The higher the score, the better the quality of life.
EPIC-26 score | over the 48 months
  urinary function will be assessed using the EPIC-26 (The Expanded Prostate Cancer Index Composite) questionnaire.
  The EPIC-26 is a self-reported scale health-related quality of life questionnaire for prostate cancer patients . It is composed of 26 items in 4 different domains: urinary incontinence, urinary irritation/obstruction, bowel, sexual, and vitality/hormonal.
  Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale. Each items as a standardized value from 0 to 100. Then the average of the standardized value is determined in each domain to crate the summary score. The higher the score, the better the quality of life.
IPSS score | over the 48 months
  urinary function will be assessed using the IPSS (International Prostate Score Symptom) questionnaire.
  The IPSS questionnaire is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35. The score is then categorized as follow: Mild (symptoms score less than or equal to 7), Moderate (symptom score range 8-19), Severe (symptom score range 20-35). The higher the score, the worse the symptoms.
IIEF-5 score | over the 48 months
  Sexual function will be assessed using the IIEF-5 (The International Index of Erectile Function) questionnaire.
  The IIEF-5 Questionnaire is composed of 5 items with 5 possible answers rating from 1 to 5 (very low, low, moderate, high, very high).
  The score is the sum of the ordinal responses to the 56 items. It is then categorized as follow: 22-25: No erectile dysfunction, 17-21: Mild erectile dysfunction, 12-16: Mild to moderate erectile dysfunction, 8-11: Moderate erectile dysfunction, 5-7: Severe erectile dysfunction. The higher the score, the better the sexual function.
patient proportion with controlled disease (Control of the pathology) | 48 months
  The main objective is the estimation of FOCAL HIFU treatment efficacy defined as the percentage of positive biopsies in the treated lobe at 48 months after inclusion.
Ancillary study: Measure of anti-tumoral immunity induction | over the 48 months
  The consequences of HIFU treatment over immune anti-tumoral induction will be estimated by the description of Programmed death-ligand 1/ligand 2 (PDL1/L2) overexpression on immune cells and overexpression of Programmed cell death 1 (PD-1) on T lymphocytes (T-cells).
Ancillary study: Measure of Circulating Tumor Cells (CTC) number reduction | over the 48 months
  The consequences of HIFU treatment over Messenger RNA (mRNA) will be estimated by measure of CTC number reduction.
Ancillary study: Measure of ncRNA (non-coding RNA) PCA3 (Prostate cancer gene 3) level reduction. | over the 48 months
  The consequences of HIFU treatment over PCA3 will be estimated by measure of ncRNA PCA3 level reduction.

CONTACTS AND LOCATIONS:
Locations (15):
- France (14):
  - Polyclinique du parc Rambot, Aix-en-Provence
  - Clinique Saint-Vincent, Besançon
  - Service d'Urologie, Clinique Tivoli Ducos, Bordeaux
  - Groupe Hospitalier Pellegrin - CHU, Bordeaux
  - Hôpital L. Pasteur, Hôpitaux Civils de Colmar, Colmar
  - Service d'Urologie CHRU de Lille, Hôpital HURIEZ, Lille
  - Service d'Urologie Générale de Santé - Hôpital Privé La Louvière, Lille
  - Service d'Urologie et Chirurgie de la Transplantation, Hôpital Edouard Herriot,, Lyon
  - Service d'urologie Assistance Publique - Hôpitaux de Marseille - Hôpital Marseille Nord, Marseille
  - Département d'Urologie, Institut Montsouris, Paris
  - Centre Hospitalier Lyon Sud - Hospices Civils de Lyon, Pierre-Bénite
  - Clinique Urologique Nantes Atlantis, Saint-Herblain
  - Service d'Urologie, Hôpital Foch, Suresnes
  - CHU de Toulouse - Hôpital de Rangueil, Toulouse
- Clinique Générale Beaulieu - Swiss International Prostate Center, Geneva, Sweden

REFERENCES:
- See also: Related Info — http://www.rhu-perfuse.fr/homepage/WP1-clinique.html